CLINICAL TRIAL: NCT01700166
Title: Safety of Autologous Human Umbilical Cord Blood in the Treatment of Stroke in Children.
Brief Title: Umbilical Cord Blood in the Treatment of Stroke in Children.
Acronym: Pedi Stroke
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator relocated; Study may resume in Fl Hosp. for Children, Orlando FL
Sponsor: Aryn Knight (Other)
Collaborators: The Institute for Rehabilitaion and Research Foundation (Other); Cord Blood Registry, Inc. (Industry); The University of Texas Health Science Center, Houston (Other); M.D. Anderson Cancer Center - Houston (Unknown); Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Aryn Knight, AVP Research, Memorial Hermann Health System
Organization: Memorial Hermann Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JB IND #14576
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Arterial Ischemic Stroke (AIS) in Children
Keywords: Autologous; Cord Blood; Stem Cells; Pediatric stroke; Children with ischemic stroke; Cerebral Palsy; Perinatal AIS
MeSH Terms: conditions — Ischemic Stroke; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biologic; Cord Blood Stem Cells; Intravenous injection (Experimental): Autologous Human Umbilical Cord Blood derived Stem Cell injection
  Interventions: Biological: Autologous Human Cord Blood derived Stem Cell injection

INTERVENTIONS:
Biological: Autologous Human Cord Blood derived Stem Cell injection — One time intravenous (in the vein) injection with two year follow-up
  Other Names: Patient's own cord blood; Patient's own stem cells

SUMMARY:
The specific aims of this study are:

1. To determine if Human Umbilical Cord Blood (hUCB) infusion is safe in children with perinatal arterial ischemic stroke (AIS).
2. To determine if late functional outcome, physiologic response, and anatomic findings are changed following hUCB infusion in children with perinatal AIS.

DETAILED DESCRIPTION:
This study will enroll ten pediatric patients who have their umbilical cord blood banked with Cord Blood Registry, Inc. (CBR), who have been diagnosed with an arterial ischemic stroke (AIS), and whose caregivers contacted CBR, Inc. to notify them that the child has experienced an AIS around the time of birth.

After receiving permission to release the patient's contact information, the CBR team will then relay the contact information to the Stem Cell Study Group at the University of Texas - Houston (UT) / Children's Memorial Hermann Hospital (CMHH) who will contact the family, explain the study, and send a consent form for their review.

Several weeks prior to the scheduled procedure date, the patient will go to their family doctor for a physical evaluation and have blood drawn to rule out problems with the child's health.

After successfully meeting initial pre-screening criteria, the patient's family will make their own arrangements to travel to Houston for the study procedures.

Once the patient is in Houston, he/she will undergo baseline assessments, including physical, neurological exams and tests, speech therapy testing, laboratory tests, and imaging (MRI) of the brain. If any of the blood tests are abnormal, or the patient has an active infection, the procedure may be postponed or the patient may possibly be excluded from the study.

If the patient continues to meet all criteria, the frozen cord blood will be shipped overnight to a special lab in Houston, TX for processing. Once release criteria have been met, the cells will be brought to the CMHH for infusion into the patient's vein. The patient will remain at CHMM for 24 hours of monitoring, after which they will be allowed to go home. Patients will be called daily by the research staff through Day 14, and once a month after that.

Patients will return to Houston, Texas for 6 month, 1 year and 2 year follow-up visits for repeat assessments, tests, and exams just like at the baseline visit. The MRI of the brain will only be repeated at the 6 month visit.

ELIGIBILITY:
Inclusion Criteria:

1. Between 6 weeks and 6 years of age on the day of study cord blood infusion.
2. MRI documented single arterial distribution infarction.
3. Initial injury occurring in the pre-natal or perinatal period.
4. Ability of caregivers to understand and speak English
5. Ability of child and caregiver to travel to Houston, and stay for at least 4 days, and to return for all Follow-up visits (patient is responsible for cost of travel and lodging while in Houston)

Exclusion Criteria:

Inability to obtain all pertinent medical records, including pertinent physician notes, laboratory findings, and radiographic images, related to the original injury, hospitalization and rehabilitation - must be sent to research team at least 14 days prior to scheduled study cord blood treatment.

1. Recent radiographic evidence (imaging performed within past 2 weeks) of extensive stroke as evidenced by >100ml lesion.
2. Multifocal infarctions on screening MRI.
3. Evidence of hypoxic-ischemic encephalopathy on screening MRI.
4. Uncorrected coagulopathy during the baseline period defined as INR > 1.4; PTT> 35 sec; PLT < 100,000.
5. Known history of:

   1. Recently diagnosed infection (within past 2 weeks) requiring treatment and/or medical intervention.
   2. Renal disease or altered renal function as defined by serum creatinine > 1.5 mg/dL at admission.
   3. Hepatic disease or altered liver function as defined by SGPT > 150 U/L, and/or T. Bilirubin >1.3 mg/dL at enrollment.
   4. Malignancy.
   5. Immunosuppression as defined by WBC < 3 (10x3) at admission.
   6. HIV, Hepatitis B, Hepatitis C.
6. Pneumonia, or chronic lung disease requiring oxygen.
7. Cord blood sample contamination.
8. Participation in a concurrent intervention study.
9. Desire for organ-donation in the event of death.
10. Unwillingness or inability to stay for at least four days following cord blood infusion (should any problems arise following the infusion) and to return for 6 month, 1 year, and 2 year follow-up visits.

Ages: 6 Weeks to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome measure | Two years
  Physiological (e.g., SSEP, EEG) and anatomic outcome (MRI) changes will be evaluated by repeating assessments, clinical tests and imaging exams at the pre-treatment and follow-up visits.

SECONDARY OUTCOMES:
Speech Therapy Specific Neuropsychological outcome measures | Two years
  Age appropriate Neurologic examinations and speech therapy specific standardized testing will be performed pre-treatment and at all follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy C. Foster, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Linda S. Baumgartner, MS, CCC-SLP, LSLS, Cert.AVT, Principal Investigator — Florida Hospital for Children - Orlando; James E. Baumgartner, MD, Study Chair — Florida Hospital for Children - Orlando
Locations (1):
- Children's Memorial Hermann Hospital; University of Texas Health Science Center - Houston, Houston, Texas, United States